CLINICAL TRIAL: NCT03233360
Title: Hepatocellular Carcinoma Registry in Asia: The INSIGHT Registry
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Asia-Pacific Hepatocellular Carcinoma (AHCC) Trials Group (Unknown); Singapore Clinical Research Institute (Other); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AHCC08 INSIGHT
Record Dates: First submitted 2017-07-18; First posted 2017-07-28 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The INSIGHT ('Insight into Real-world Practice of Management of HCC in Asia-Pacific') registry is designed as a multi-centre longitudinal cohort study of patients diagnosed with HCC between 1st January 2013 and 31st December 2019 in nine countries (i.e., South Korea, Taiwan, Thailand, Japan, China, Hong Kong, Australia, New Zealand and Singapore). Approximately 30% of the sample size will be identified retrospectively and 70% will be identified prospectively from the start date of the registry (October 2016), with an even distribution of consecutively diagnosed patients within the different years.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged 21 or above.
* Patient with confirmed diagnosis of HCC between 1st January 2013 and 31st December 2019 based on one or more of the following criteria:

  * American Association for the Study of Liver Diseases (AASLD) criteria
  * Asian Pacific Association for the Study of the Liver (APASL) criteria
  * Histology/cytology
  * Space occupying lesion in the liver and an serum alpha-feto protein of > 400 ng/mL in a patient with chronic viral hepatitis or cirrhosis from any cause
* Informed consent form (ICF) to be presented and signed by patients who are still alive at the point of study enrolment, per local regulations. For the collection of data for deceased subjects, appropriate waiver of consent as per local regulations and guidelines will have to be in place.
* Patient who is being followed-up at the participating site.

Exclusion Criteria:

- Patients participating in any HCC-related therapeutic/interventional clinical trial.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HCC between 1st January 2013 and 31st December 2019 in nine countries (i.e., South Korea, Taiwan, Thailand, Japan, China, Hong Kong, Australia, New Zealand and Singapore).
Sampling Method: Non-Probability Sample
Enrollment: 2533 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From diagnosis or treatment initiation to date of death due to any cause, or last known vital status date, up to 2 years
Progression-free survival | From treatment initiation for advanced or metastatic HCC to the first date of disease progression or death due to any cause, whichever occurred first, up to 2 years
  Patients lost for follow up or withdrawn from the study will be censored at the last disease assessment date
Time to progression | From the start of treatment for a disease until disease progression, up to 2 years
  Measuring the time to progression is one way to see how well a new treatment works. Also called TTP.
Overall Survival Rate | 5 years from date of diagnosis
  The percentage of people in a study or treatment group who are still alive for a certain period of time after they were diagnosed with or started treatment for a disease, such as cancer. The overall survival rate is often stated as a five-year survival rate, which is the percentage of people in a study or treatment group who are alive five years after their diagnosis or the start of treatment. Also called survival rate.
Best Overall Response Rate (BORR) | From treatment initiation to CR or PR, up to 2 years
  The proportion of patients who had either a complete response (CR) or partial response (PR) after initiation of treatment for HCC
Disease Control Rate (DCR) | From treatment initiation to SD, CR or PR, up to 2 years
  The proportion of patients who had either stable disease (SD) for ≥ 6 months, a CR or PR after initiation of treatment for HCC
Disease Free Survival (DFS) | From the time from completing adjuvant/neoadjuvant treatment to the date of HCC recurrence, or the date of death due to any cause, whichever occurred first, up to 2 years
  Patients lost for follow up will be censored at the last disease assessment date; DFS rate at 2 years - defined as the proportion of HCC patients who are alive and cancer free 2 years after completion of adjuvant/neoadjuvant treatment
Recurrence rate | From the time from a CR to treatment to the first recurrence of HCC, up to 2 years
  The proportion of patients who experience a recurrence of HCC after having had a CR to treatment
Sites of recurrence | From the time from a CR to treatment to the first recurrence of HCC, up to 2 years
  local/ regional / distant; specify site(s)
Time to treatment recurrence | From the time from a CR to treatment to the first recurrence of HCC, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (34):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
- China (6):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Southwest Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Guangxi Medical University Cancer Center, Nanning, Guangxi
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Queen Mary Hospital, Hong Kong, Hong Kong
- Japan (4):
  - Kinki University School of Medicine, Ōsakasayama, Osaka
  - National Cancer Centre, Japan, Chūōku, Tokyo
  - Kyorin University School of Medicine, Mitaka-shi, Tokyo
  - University of Tokyo, Tokyo
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (8):
  - St Vincent Hospital, Catholic University Medical College, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Asan Medical Centre, Seoul
  - St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital-KS, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (3):
  - Chulabhorn Hospital, Bang Khen, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - National Cancer Institute, Ratchathewi, Bangkok

IPD SHARING:
Plan to Share IPD: No